CLINICAL TRIAL: NCT06313593
Title: A Phase 1, Open-Label, Multicenter Study of INCB160058 in Participants With Myeloproliferative Neoplasms
Brief Title: A Study to Evaluate the Safety, Tolerability of INCB160058 in Participants With Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB160058-101; 2024-520353-21-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Myeloproliferative Neoplasms
Keywords: Myeloproliferative Neoplasms; INCB160058; Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Dose Escalation - with MF, PV or ET (Experimental): INCB160058 will be administered at a protocol defined starting regimen to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myelofibrosis (MF), polycythemia vera (PV) or essential thrombocythemia (ET) will enroll in this group.
  Interventions: Drug: INCB160058
- Part 1 Dose Escalation - with MF SubOpt R (Experimental): INCB160058 will be administered at a protocol defined starting regimen and will allow for the evaluation of INCB160058 in combination with a standard disease-directed therapy to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myelofibrosis (MF), suboptimal response to a standard disease-directed therapy (SubOpt R) will enroll in this group.
  Interventions: Drug: INCB160058; Drug: Standard disease-directed therapy
- Part 2 Dose Expansion - with MF, PV or ET (Experimental): INCB160058 will be administered at the RDE(s) identified during Part 1. Participants with MF, PV or ET will enroll in this group.
  Interventions: Drug: INCB160058
- Part 2 Dose Expansion - with MF SubOpt R (Experimental): INCB160058 will be administered as an add-on therapy in combination with a standard disease-directed therapy at the RDE(s) identified during Part 1. Participants with myelofibrosis (MF), suboptimal response to a standard disease-directed therapy (SubOpt R) will enroll in this group.
  Interventions: Drug: INCB160058; Drug: Standard disease-directed therapy

INTERVENTIONS:
Drug: INCB160058 — Oral; Tablet
Drug: Standard disease-directed therapy — A standard disease-directed therapy will be administered according to Prescribing Information/SmPC.
  Arms: Part 1 Dose Escalation - with MF SubOpt R; Part 2 Dose Expansion - with MF SubOpt R

SUMMARY:
This study is being conducted to assess the Safety, Tolerability, and Pharmacokinetics of INCB160058 in Participants With Myeloproliferative Neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* MF:

  * Intermediate-1 or higher risk PMF, post-PV MF, or post-ET MF with evidence of minimum burden of disease based on splenomegaly, and for the monotherapy cohort, participants must have been previously treated with at least 1 JAK inhibitor for ≥ 12 weeks and resistant, refractory, intolerant to, or have lost response to JAK inhibitor treatment.
  * For the MF SubOpt R cohort: Therapeutic regimen prior to enrollment as defined in the protocol and unlikely to benefit from further monotherapy in the opinion of the investigator.
* PV: Confirmed diagnosis of PV and previously treated with at least 1 prior standard cytoreductive therapy and are resistant, refractory, intolerant to, or have lost response to treatment.
* ET: Confirmed diagnosis of high-risk ET as defined in the protocol and previously treated with at least 1 prior standard cytoreductive therapy and are resistant, refractory, intolerant to, or have lost response to treatment.
* Life expectancy > 6 months.
* Willingness to undergo a pretreatment and regular on-study bone marrow biopsies and aspirations (as appropriate to disease).
* Existing documentation of JAK2V617F mutation from a qualified local laboratory.

Exclusion Criteria:

* Presence of a hematological malignancy requiring treatment, other than PMF, post-PV MF, post-ET MF, PV, or ET.
* Prior history of major bleeding or thrombosis within the 3 months prior to study enrollment.
* Participants with abnormal hematologic, hepatic, or renal function based on laboratory evaluation.
* Has undergone prior allogenic or autologous stem-cell transplantation or allogenic stem-cell transplantation is planned
* Active invasive malignancy.
* Significant concurrent, uncontrolled medical condition.
* Acute or chronic HBV, active HCV or known HIV.
* Any prior MPN-directed therapy within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* Participants undergoing treatment with G-CSF or GM-CSF, romiplostim, or eltrombopag at any time within 4 weeks before the first dose of study treatment.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2028-10-09 (Estimated); Study Completion 2028-10-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Number of participants with TEAEs leading to dose modification or discontinuation | Up to 2 years and 30 days
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
INCB160058 and a standard disease-directed therapy pharmacokinetic (PK) in Plasma | Up to Day 57
  INCB160058 and the protocol defined standard disease-directed therapy concentration in plasma.
For participants with MF: Response using the revised IWG-MRT and ELN response criteria for MF | Week 12 and 24 and then every 24 weeks up to 2 years
  Defined as the percentage of participants with Response using the revised International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) response criteria.
For participants with MF: Percentage of participants achieving spleen volume reduction as defined in the protocol | Week 12 and Week 24
  Defined as percentage of participants with a protocol defined Spleen Volume Reduction.
For participants with PV: Response using revised IWG-MRT and ELN response criteria for PV | Week 12 and 24 and then every 24 weeks up to 2 years
  Defined as the percentage of participants with Response using the revised International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) response criteria.
For participants with ET: Response using revised IWG-MRT and ELN response criteria for ET | Week 12 and 24 and then every 24 weeks up to 2 years
  Defined as the percentage of participants with Response using the revised International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) response criteria.
For all participants: Percentage of participants achieving ≥ 50% reduction from baseline of total symptom score (TSS) | Week 24
  Defined as the percentage of participants achieving ≥ 50% reduction from baseline of TSS.
For all participants: Symptom improvement in TSS at Weeks 12 and 24 relative to baseline as measured by the Myeloproliferative Neoplasms Symptom Assessment Form (MPN-SAF) TSS. | Week 12 and Week 24
  Defined as the proportion of participants who achieve a protocol defined reduction in Total Symptomatic Score (TSS) relative to baseline as measured by the MPN-SAF TSS.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical, Study Director — Incyte Corporation
Locations (31):
- United States (14):
  - The University of Alabama At Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - The University of Kansas Cancer Center Kucc University of Kansas Clinical Research Center, Fairway, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Cornell Medical Center, New York, New York
  - Sloan Kettering Institute For Cancer Research, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Qc, Montreal, Quebec
  - McGill University Jewish General Hospital, Montreal, Quebec
- France (2):
  - Hospital Saint Louis, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - University Medical Center Rwth Aachen, Aachen
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Halle (Saale), Halle
- Italy (3):
  - Aou Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Universitatsspital Zurich, Zurich
- United Kingdom (2):
  - Guys and St Thomas Nhs Foundation Trust, London
  - Genesiscare Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate the Safety, Tolerability of INCB160058 in Participants With Myeloproliferative Neoplasms — https://www.incyteclinicaltrials.com/study/?id=INCB160058-101&SearchTerm=INCB160058-101&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=